CLINICAL TRIAL: NCT01529086
Title: Determining the Likelihood of Prostate Cancer Detection in Men Taking Dutasteride When Biopsy is Performed 'for Cause'.
Brief Title: For Cause Prostate Biopsy in REDUCE Population Trial
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Stephen Jones, Chairman of Department of Regional Urology, The Cleveland Clinic
Other Study IDs: REDUCE-FOR CAUSE; 115686 (Other: GSK)
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; dutasteride; for cause prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Subjects on Dutasteride that meet the following criteria:
  1. . A rise in PSA from nadir at any time post-nadir
  2. . PSA change from baselin >0.2 mg/ml at any time post-baseline
  3. . Abnormal DRE at any time post-baseline
  4. . Free-PSA <12% at any time post-baseline
  5. . At least one of the above 4 criteria
  6. Subjects on Dutasteride that do not meet the above criteria
- Group 2: Subjects on placebo treatment that meet the following criteria:
  1. Change from baseline PSA between 0.0 and 0.35 (ie, 0.0 ≤ change from baseline PSA < 0.35) at any time post-baseline. Note that in REDUCE PSA was recorded to the nearest 0.1.
  2. Abnormal DRE at any time post-baseline
  3. Change from baseline PSA ≥ 0.35 at any time post-baseline
  4. Change from baseline PSA ≥ 0.75 at any time post-baseline
  5. PSA ≥ 2.5 at any time post-baseline
  6. PSA ≥ 4.0 at any time post-baseline
  7. Percent Free PSA < 12% at any time post-baseline
  8. At least one of the above 7 criteria.
  9. Subjects on placebo that do not meet the above criteria

SUMMARY:
The REDUCE trial was conducted to determine whether dutasteride reduces the risk of incident prostate cancer, as detected on biopsy, among men who are at increased risk for the disease. Dutasteride was compared with placebo for 4 years period. Results showed a relative risk reduction of 22.8 % (95% CI: 15.2 to 29.8)in prostate cancer.

For REDUCE, biopsies were defined as "protocol biopsy" if performed at certain timeframes, and "for cause" if outside these predetermined timeframes.

The investigators propose a post hoc analysis that would allow them to include biopsies that really justified a clinical indication, but were excluded from "for cause" analysis based on occurring at either the 2 or 4 year timeframes.

Thus the investigators propose analysis of both REDUCE groups by every yearly timeframe as:

Group 1--dutasteride group biopsied "for cause" using several definitions: biopsy of patients who received dutasteride whose PSA rose from nadir as defined in your own protocol,who had a PSA rise>0.2 ng/ml or who had a new abnormal DRE or had a free PSA<12% . The investigators define these as such because this would reasonably instigate biopsy if the clinician had a patient with this scenario in the non-study setting.

Group 2--placebo group biopsied "for cause" using several definitions, regardless of timeframe but reported at each year of the study and aggregate, with the aggregate number being the primary outcome. Thus the investigators would request results of biopsy of patients who received placebo To establish differences in biopsy positive rates the groups as per each definition listed, to determine if dutasteride decreased the likelihood of "for cause" biopsy compared to "not for cause" biopsy, and if there is a difference in cancer detection risk rate depending on cause vs. no cause in that group compared to placebo.

DETAILED DESCRIPTION:
Purpose: Determining the likelihood of prostate cancer detection in men taking dutasteride when biopsy is performed 'for cause'.

Population: The population of interest is the REDUCE Biopsied population, that is, all subjects in the Efficacy population who have at least one post-baseline biopsy reviewed by the Central Pathology Laboratory.

Analyses: Initial interest will be focused on data from the Year 1-2 time period, to avoid the potential effect of the cancer diagnoses from the Year 2 scheduled biopsies on the assessments utilized in the "for cause" definitions. Only PSA data from Years 1-2 and baseline will be utilized in the computation of the various PSA metrics, and only Central Pathology results from Years 1-2 will be utilized to establish post-baseline diagnoses. PSA values on or within 42 days after date of biopsy will be excluded from the analyses, to avoid potential effects of biopsy on the PSA value.

For each of the 2 groups of subjects, the following will be summarized: number of subjects meeting the corresponding criteria, number and % of subjects diagnosed with prostate cancer, number and % of such subjects diagnosed with Gleason 7-10, and number and % of subjects diagnosed with either prostate cancer, HGPIN or ASAP. Summaries of the numbers of subjects meeting each of the specific criteria for group 1 (a through e) and Group 2 (a through h) will be provided.

In addition, summaries investigating the effect of baseline variables (such as age, family history of prostate cancer, prostate volume, percent free PSA, number of cores at the entry biopsy) on the occurrence of prostate cancer diagnoses and Gleason 7-10 diagnoses may be developed.

ELIGIBILITY:
Inclusion Criteria:

Group 1-subjects in the dutasteride treatment group who meet the following sets of criteria:

* A rise in PSA from nadir at any time post-nadir
* PSA change from baseline >0.2 ng/ml at any time post-baseline
* Abnormal DRE at any time post-baseline
* Free PSA<12% at any time post-baseline
* At least one of the above 4 criteria.

Group 2-subjects in the placebo treatment group who meet the following sets of criteria:

* Change from baseline PSA between 0.0 and 0.35 (ie, 0.0 ≤ change from baseline PSA < 0.35) at any time post-baseline. Note that in REDUCE PSA was recorded to the nearest 0.1.
* Abnormal DRE at any time post-baseline
* Change from baseline PSA ≥ 0.35 at any time post-baseline
* Change from baseline PSA ≥ 0.75 at any time post-baseline
* PSA ≥ 2.5 at any time post-baseline
* PSA ≥ 4.0 at any time post-baseline
* Percent Free PSA < 12% at any time post-baseline
* At least one of the above 7 criteria.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: REDUCE trial participants
Sampling Method: Probability Sample
Enrollment: 6608 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cancer detection risk among the groups in the "for cause" context | 4 years
  Determination of differences in cancer detection risk rate depending on cause vs no cause in that group compared to placebo

SECONDARY OUTCOMES:
Dutasteride as a key factor in the likelihood of "for cause" biopsy | 4 years
  Determination of dutasteride as an item in decreasing the likelihood of "for cause" biopsy compared to "not for cause" biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Jones, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andriole GL, Bostwick DG, Brawley OW, Gomella LG, Marberger M, Montorsi F, Pettaway CA, Tammela TL, Teloken C, Tindall DJ, Somerville MC, Wilson TH, Fowler IL, Rittmaster RS; REDUCE Study Group. Effect of dutasteride on the risk of prostate cancer. N Engl J Med. 2010 Apr 1;362(13):1192-202. doi: 10.1056/NEJMoa0908127. PMID 20357281